CLINICAL TRIAL: NCT04131192
Title: A Phase Ib, Multi-center, Open-label Study of Z650 and Gemcitabine in Advanced Pancreatic Cancer
Brief Title: Gemcitabine and Z650 in Treating Patients With Metastatic or Recurrent Pancreatic Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Combined with the analysis of the existing data of the trial, there was no obvious advantage compared with the clinical standard treatments, and the clinical trial was decided to be terminated based on the benefit of the subjects.
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCD-DZ650-19-001
Record Dates: First submitted 2019-10-10; First posted 2019-10-18 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- z650 and Gemcitabine (Experimental): Z650:250 or 300 or 200 mg/d, starting on the 2nd day, once a day, continuous administration, or about half an hour after a meal Gemcitabine: intravenously at 1000 mg/m2 on Days 1, 8, of a 21-day cycle FOR the 4-6 cycles
  Interventions: Drug: Z650; Drug: Gemcitabine

INTERVENTIONS:
Drug: Z650 — 250 or 300 or 200 mg/d, starting on the 2nd day, once a day, continuous administration, or about half an hour after a meal
  Other Names: larotinib
Drug: Gemcitabine — Gemcitabine will be administered intravenously at 1000 mg/m2 on Days 1, 8, of a 21-day cycle ，for 4-6 cycles
  Other Names: Gemzar

SUMMARY:
This phase IB trial is studying how well giving gemcitabine together with Z650 works in treating patients with metastatic or recurrent pancreatic cancer.

DETAILED DESCRIPTION:
This phase IB trial is studying how well giving gemcitabine together with Z650 works in treating patients with metastatic or recurrent pancreatic cancer.This phase IB trial is Multi-center and open。

ELIGIBILITY:
Inclusion Criteria:

18 ≤ age ≤ 75 years old, male or female is not limited; Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1 Life expectancy of ≥ 12 weeks Pathologically confirmed advanced pancreatic cancer defined as non-operable in a curative intent, locally recurrent, or metastatic disease.

Exclusion Criteria:

adjuvant treatment with gemcitabine within 6 months prior to the first dose; Radiotherapy and anti-cancer Chinese patent medicine treatment were performed within 4 weeks before the first dose; Gastrointestinal diseases that could affect the absorption of Z650, (e.g., serious swallowing obstruction, chronic diarrhea, bowel obstruction); Doppler ultrasound evaluation of Left ventricular ejection fraction < 50%

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2021-09-09 (Actual); Study Completion 2021-09-09 (Actual)

PRIMARY OUTCOMES:
Rate of dose limiting toxicities of each subject | 21 days
  Rate will be assessed through summaries of adverse events, clinical laboratory abnormalities, and changes in physical exam and vital signs. All subjects who receive a single dose of study medication will be considered evaluable for safety.

SECONDARY OUTCOMES:
Adverse events related to pulse dose Z650 and gemcitabine | up to 4 weeks after last dose
  description, timing, grade (Common Terminology Criteria for Adverse Events Version 5.0 [CTCAE v5.0]), severity, seriousness, and relatedness
Overall response rate (ORR) | up to approximately 24 months
  Overall response rate (ORR), defined as a partial response (PR) or complete response (CR) occurring at any point post-treatment according to Response Evaluation Criteria in Solid Tumors as assessed by RECIST v1.1
Disease Control Rate (DCR) | up to approximately 24 months
  DCR, proportion of patients with best overall response of CR, PR or stable disease (SD)
Duration of Response (DOR) | up to approximately 24 months
  DOR, defined as time from the first documented CR or PR to first documented progression or death due to any cause
Progression-free Survival (PFS) | up to approximately 24 months
  PFS, defined as time from date of treatment to disease progression or death due to any cause
Overall Survival (OS) | up to approximately 24 months
  OS, defined as time from date of treatment to death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: shu zhang, Principal Investigator — Shandong Cancer Hospital and Institute; lianke liu, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (2):
- China (2):
  - Jiangsu Province Hospital, Nanjing, China/jiangsu
  - shandong Cancer Hospital, Jinan, China/shandong

IPD SHARING:
Plan to Share IPD: No